CLINICAL TRIAL: NCT02891434
Title: Analysis of Interaction of Different Devices in a Virtual Reality Task in Patients With Duchenne Muscular Dystrophy
Brief Title: Analysis of a Virtual Reality Task in Patients With Duchenne Muscular Dystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carlos Bandeira de Mello Monteiro, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 248/15
Record Dates: First submitted 2016-08-17; First posted 2016-09-07 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; motor learning; motor abilities
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Acquisition on TouchScreen (Experimental): Subjects practice the task and retention TouchScreen, transfer 1 on LeapMotion and transfer 2 on Kinect
  Interventions: Device: Acquisition on TouchScreen
- Acquisition on Kinect (Experimental): Subjects practice the task and retention Kinect, transfer 1 on TouchScreen and transfer 2 on LeapMotion.
  Interventions: Device: Acquisition on Kinect
- Acquisition on LeapMotion (Experimental): Subjects practice the task and retention LeapMotion, transfer 1 on TouchScreen and transfer 2 on Kinect.
  Interventions: Device: Acquisition on LeapMotion
- Acquisition on TouchScreen Control Group (Active Comparator): Subjects practice the task and retention TouchScreen, transfer 1 on LeapMotion and transfer 2 on Kinect
  Interventions: Device: Acquisition on TouchScreen
- Acquisition on Kinect Control Group (Active Comparator): Subjects practice the task and retention Kinect, transfer 1 on TouchScreen and transfer 2 on LeapMotion.
  Interventions: Device: Acquisition on Kinect
- Acquisition on LeapMotion Control Group (Active Comparator): Subjects practice the task and retention LeapMotion, transfer 1 on TouchScreen and transfer 2 on Kinect.
  Interventions: Device: Acquisition on LeapMotion

INTERVENTIONS:
Device: Acquisition on TouchScreen — Participants performed acquisition and retention on TouchScreen, transfer 1 on Kinect and transfer 2 on LeapMotion.
  Arms: Acquisition on TouchScreen; Acquisition on TouchScreen Control Group
Device: Acquisition on Kinect — Participants performed acquisition and retention on Kinect, transfer 1 on TouchScreen and transfer 2 on LeapMotion.
  Arms: Acquisition on Kinect; Acquisition on Kinect Control Group
Device: Acquisition on LeapMotion — Participants performed acquisition and retention on LeapMotion, transfer 1 on TouchScreen and transfer 2 on Kinect.
  Arms: Acquisition on LeapMotion; Acquisition on LeapMotion Control Group

SUMMARY:
The task consists in reach as much bubbles as they can, the bubbles appear on the screen of the computer and should be reached in 10 seconds. To accomplish that, three different devices will be used: (1) Kinect for Windows Microsoft - which consists of a sensor that captures body movements (including upper limbs). And (2) the Leap Motion (LMCH, Leap Motion, Inc., San Francisco, CA, USA), and (3) Touch Screen. To describe motor impairments was used the Motor Function Measure Scale; Scale Vignos and Scale Egen Klassifikation;

DETAILED DESCRIPTION:
To evaluate the performance of interaction devices was used a computer game proposed by the Department of Information Systems, University of São Paulo. Chosen due to its low cognitive demands, ease and adaptability for use in people with DMD. The program, offers a task designed to measure various neuropsychological aspects of planning, execution, spatial organization, which involves the operation of the intention to move to achieve a virtual object and the planning of this action.

Considering different interfaces, opted for three interfaces. Two of theme without physical contact, represented by (1) Kinect for Windows Microsoft - which consists of a sensor that captures body movements (including upper limbs). And (2) the Leap Motion (LMCH, Leap Motion, Inc., San Francisco, CA, USA) - virtual interface by means of a sensor, in which there is also no need to touch or physical contact , but its catchment area is focused only on hands and fingers. In addition, an interface that required physical contact -Touch Screen - a sensitive monitor to touch the computer screen itself. The use of interfaces with and without physical contact are interesting to identify the functionality of the devices.

Therefore, the game presented 126 bubbles arranged in rows and columns . The goal was that the participant could achieve (changing color) the largest number of bubbles during 10 seconds, thereby defining a range zone for the specified time.

After defining the scope zone, the therapist established a red target bubble, which was chosen in the center of bottom of range line. The participant should play this target bubble using one of the devices, Touch Screen, Kinect and Leap Motion. After touch of target bubble, the game had another red bubble in a random position, within range of area. After reaching the random bubble, the bubble target was displayed again, and so on. The game features red bubbles within the range area, and sometimes out of range, thus creating a higher degree of difficulty and to encourage participants to challenge their limits.

The Participants were divided into groups which performed the tasks with different interaction devices, more virtual feature (not touch the computer using Kinect or leap motion) or real (to touch the computer screen).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of DMD.

Exclusion Criteria:

* presence disorders in cognitive function that would prevent comprehension of the experimental instruction.

Ages: 9 Years to 34 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Motor performance improvement in a virtual Timing Coincident task, with better performance on the LeapMotion compared to TouchScreen and Kinect. | 3 months
  Analysis of the motor performance using a virtual Coincident timing task in different devices to compare wether a task with or without contact promote better performance for people with Duchenne Muscular Dystrophy

CONTACTS AND LOCATIONS:
Overall Officials: Carlos BM Monteiro, Ph.D., Principal Investigator — University of Sao Paulo
Locations (1):
- Escola de Artes,Ciencias e Humanidades da Universidade d Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Freitas BL, da Silva TD, Crocetta TB, Massetti T, de Araujo LV, Coe S, Dawes H, Caromano FA, Monteiro CBM. Analysis of Different Device Interactions in a Virtual Reality Task in Individuals With Duchenne Muscular Dystrophy-A Randomized Controlled Trial. Front Neurol. 2019 Jan 29;10:24. doi: 10.3389/fneur.2019.00024. eCollection 2019. PMID 30761066